CLINICAL TRIAL: NCT04792203
Title: The Evaluation of the Ultrasound-guided Clinical Procedure Simulation Curriculum
Status: Active, not recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202011111RIND
Record Dates: First submitted 2021-03-07; First posted 2021-03-10 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Ultrasound Performance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Ultrasound is a non-radiated diagnostic tool that can be performed at the bedside in emergency departments and critical care settings. Traditionally, junior residents learn from patients by performing sonography on them. However, patient rights, patient safety, and medical quality are raising concerns.

How to enable junior doctors to be effectively familiar with ultrasound operations and to effectively integrate them into daily practice has become a major challenge in medical education. Also, the ultrasound-guided clinical procedure is included in the ultrasound core applications in the American College of Emergency Physicians statements.

This aim of this study is to establish an ultrasound-guided simulation curriculum and to evaluate the efficacy. The subjects of the study are junior doctors who are interested in clinical procedures in the emergency department or other relevant medical departments, and it is estimated that 200 people will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* participants attended the curriculum.

Exclusion Criteria:

* not attended the curriculum

Min Age: 25 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: inexperience doctors including the 1st-3rd post-graduate year residents
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ultrasound-guided clinical procedure | 3 months
  thoracocentesis, abdominal tapping, vasculizastion

CONTACTS AND LOCATIONS:
Overall Officials: WAN-CHING LIEN, Principal Investigator — NTUH
Locations (1):
- Department of Emergency Medicine, National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Huang SS, Lin CH, Lin SY, Huang CT, Lien WC. How to enhance the novices' learning in ultrasound-guided procedures utilizing handmade phantoms? BMC Med Educ. 2024 Dec 18;24(1):1444. doi: 10.1186/s12909-024-06458-z. PMID 39695599
- [Derived] Huang CT, Lin CH, Lin SY, Huang SS, Lien WC. A feasibility study of a handmade ultrasound-guided phantom for paracentesis. BMC Med Educ. 2024 Mar 29;24(1):351. doi: 10.1186/s12909-024-05339-9. PMID 38553674